CLINICAL TRIAL: NCT00132912
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of SCH 530348 in Subjects Undergoing Non-Emergent Percutaneous Coronary Intervention
Brief Title: Safety of SCH 530348 in Subjects Undergoing Non-Emergent Percutaneous Coronary Intervention (Study P03573)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P03573
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Arterial Obstructive Diseases; Coronary Disease
Keywords: Platelets; Platelet Aggregation Inhibitors; Protease-Activated Receptor 1; Hemorrhage
MeSH Terms: conditions — Arterial Occlusive Diseases; Coronary Disease; Hemorrhage | interventions — vorapaxar

INTERVENTIONS:
Drug: SCH 530348

SUMMARY:
The object of the study is to determine whether different doses of SCH 530348, when added to standard medical care in persons undergoing percutaneous coronary intervention, will increase the risk of bleeding.

A secondary objective is to determine whether patients treated with SCH 530348 have fewer cardiac events such as heart attack, bypass surgery, or death compared with those persons treated with the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* A person who is 45 years or older and is mentally competent to provide a signed written informed consent.
* A person who is scheduled to undergo a percutaneous coronary intervention or a heart catheterization with the intent to undergo a percutaneous coronary intervention.
* If a woman is of childbearing potential (ie, before menopause), she must test negative for pregnancy and agree to use a reliable method of birth control.

Exclusion Criteria:

* Pregnancy
* Recent stroke
* Active internal bleeding or a history of a bleeding disorder
* Increased risk of bleeding
* Severe high blood pressure
* Liver or kidney disease
* Low platelet count
* Condition such as alcoholism, mental illness, or drug dependence
* Ongoing chest pain
* Planned or ongoing treatment with a blood thinning medication
* A serious condition or illness that would interfere with participation in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2005-08-30 (Actual); Primary Completion 2007-01-28 (Actual); Study Completion 2007-01-28 (Actual)

PRIMARY OUTCOMES:
Incidence of bleeding through the end of treatment in subjects undergoing percutaneous coronary intervention

SECONDARY OUTCOMES:
Incidence of bleeding throughout treatment and follow-up
Incidence of death and major adverse cardiac events

REFERENCES:
- [Derived] Becker RC, Moliterno DJ, Jennings LK, Pieper KS, Pei J, Niederman A, Ziada KM, Berman G, Strony J, Joseph D, Mahaffey KW, Van de Werf F, Veltri E, Harrington RA; TRA-PCI Investigators. Safety and tolerability of SCH 530348 in patients undergoing non-urgent percutaneous coronary intervention: a randomised, double-blind, placebo-controlled phase II study. Lancet. 2009 Mar 14;373(9667):919-28. doi: 10.1016/S0140-6736(09)60230-0. PMID 19286091
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html